Official title: Impact of Plant-Based Meat Analogues Consumption on Human Health

NCT number: NCT ID not yet assigned

Document data: January 2021

## STATISTICAL ANALYSIS PLAN

All statistical tests will be performed using R (available version). Data will be analysed for normality using Shapiro–Wilk tests. Where data are normally distributed, results will be presented as mean±standard deviation (SD) and the effect of postprandial time will be analysed using a repeated measures analysis of variance (ANOVA). Where data are not normally distributed, they will be log transformed, and if normality is not achieved, analyses will be conducted using Friedman's test with Wilcoxon's signed-rank test.

The variation in maximal concentration will be calculated as the difference between the peak concentration (Cmax) and the concentration in basal (fasting) conditions (Cmax–Fasting). Area under the curve (AUC) will be calculated considering all sampling times, including the initial "0" minute sampling point. The incremental AUC ( $\Delta$ AUC0–x hours) was calculated as the total area above the baseline concentration (i.e., AUC0-x hours–(baseline concentration multiplied by x hours). The data from questionnaires will be normally distributed and hence, repeated measures ANOVA tests will be applied to assess the effect of postprandial time. To assess the effect of VM and GM on postprandial events, appropriate comparisons will be made using t-tests for parametric data or Mann-Whitney tests for non-parametric data. P values < 0.05 will be interpreted as statistically significant.